CLINICAL TRIAL: NCT04995250
Title: Effects of Corrective Exercise Training for Improving Neuropathic Pain and Function in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/1065
Record Dates: First submitted 2021-03-26; First posted 2021-08-06 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corrective exercise training for knee Osteoarthritis (Experimental)
  Interventions: Other: corrective exercise training for knee

INTERVENTIONS:
Other: corrective exercise training for knee — All patients received 12 weeks (3 days per week) physiotherapy sessions with hot pack, TENS and Ultrasound session for 10 mints and knee isometric, quad strengthening, adductor and abductor strengthening, calf stretch, hamstring stretch, Maitland mobilization, Unconventional Corrective knee exercise protocol treatment: standing on one extremity, up and down on bosu exercise, walking to lateral direction, walking to anterio-posterior direction, walking to anterio-posterior and lateral for 20 mints. Data were collected at baseline, at week 4 and at post treatment (week 12).

SUMMARY:
Patients with neuropathic pain had longer duration of symptoms increased severity of pain, functional limitation and disability as compare to the patient with general knee osteoarthritis.

Objective: To find out the effects of corrective exercise training for improving neuropathic pain and function in knee OA patients.

DETAILED DESCRIPTION:
This study was a Quasi experimental study. It was conducted at Horizon Hospital Johar Town Lahore. The study was completed in Six months. Consecutive sampling technique was used to collect the data. The sample size of 16 patients was taken in this study to find out the effects of corrective exercises training for improving neuropathic pain and function in patients with knee osteoarthritis. For descriptive analysis we used frequency, percentages and charts. For quantitative measure. Repeated Measured ANOVA was used.

ELIGIBILITY:
Inclusion Criteria:

* ACR Criteria for osteoarthritis
* Neuropathic pain
* Age over 65
* DN4 cut off value is 4/10
* Less than 30 minutes of morning stiffness
* Grade I and II
* Crepitus on active motion
* Bony tenderness
* Bony enlargement
* No palpable warmth of synovium

Exclusion Criteria:

* Knee complain that require urgent medical attention (fracture and infection)
* Diabetes mellitus
* Patients with malignancies
* Neurological disorders
* Systematic musculoskeletal diseases (Parkinson's, rheumatoid arthritis etc)
* Incapability of understanding implication of participants

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Osteoarthritis Index | 6 months
  0-100, 0 means no disability 100 means maximum disability
Numeric pain rating scale | 6 months
  0-10,no pain and the worse pain, on an 11 point scale
Douleur Neuropathique 4 Questionnaire | 6 months
  The total score is calculated as the sum of 10 items and the cut off value for the diagnosis of neuropathic pain is a total score of 4/10

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polat CS, Dogan A, Sezgin Ozcan D, Koseoglu BF, Kocer Akselim S. Is There a Possible Neuropathic Pain Component in Knee Osteoarthritis? Arch Rheumatol. 2017 Apr 24;32(4):333-338. doi: 10.5606/ArchRheumatol.2017.6006. eCollection 2017 Dec. PMID 29901006
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Knoop J, Steultjens MP, van der Leeden M, van der Esch M, Thorstensson CA, Roorda LD, Lems WF, Dekker J. Proprioception in knee osteoarthritis: a narrative review. Osteoarthritis Cartilage. 2011 Apr;19(4):381-8. doi: 10.1016/j.joca.2011.01.003. Epub 2011 Jan 18. PMID 21251988
- [Background] Takacs J, Carpenter MG, Garland SJ, Hunt MA. The role of neuromuscular changes in aging and knee osteoarthritis on dynamic postural control. Aging Dis. 2013 Jan 15;4(2):84-99. Print 2013 Apr. PMID 23696951
- [Background] Beckwee D, Vaes P, Cnudde M, Swinnen E, Bautmans I. Osteoarthritis of the knee: why does exercise work? A qualitative study of the literature. Ageing Res Rev. 2013 Jan;12(1):226-36. doi: 10.1016/j.arr.2012.09.005. Epub 2012 Sep 28. PMID 23026409
- [Background] Sazo-Rodriguez S, Mendez-Rebolledo G, Guzman-Munoz E, Rubio-Palma P. The effects of progressive neuromuscular training on postural balance and functionality in elderly patients with knee osteoarthritis: a pilot study. J Phys Ther Sci. 2017 Jul;29(7):1229-1235. doi: 10.1589/jpts.29.1229. Epub 2017 Jul 15. PMID 28744054